CLINICAL TRIAL: NCT00299702
Title: A 2-year, Prospective, Blinded-rater, Open-label, Active-controlled, Multicenter, Randomized Study of Long-term Efficacy and Effectiveness Comparing Risperdal® Consta® and Abilify® (Aripiprazole) in Adults With Schizophrenia
Brief Title: Evaluation of Effectiveness of Risperdal® Consta® Compared to Abilify® Over a Two-year Period in Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Janssen, LP (Industry)
Responsible Party: Vice President, Medical Affairs, Ortho-McNeil Janssen Scientific Affairs, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR006121; RISSCH4060 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Results first posted 2010-03-16 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Schizophrenia; Relapse; Remission; Treatment Outcome; long-acting injectable
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Recurrence | interventions — Aripiprazole; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 002 (Active Comparator)
  Interventions: Drug: Abilify
- 001 (Experimental)
  Interventions: Drug: Risperidal Consta

INTERVENTIONS:
Drug: Abilify — 10-30 mg once daily for 104 weeks
  Arms: 002
Drug: Risperidal Consta — 25mg, 37.5mg, or 50mg every 2 weeks for 104 weeks
  Arms: 001

SUMMARY:
The purpose of this study is to compare the effectiveness of two antipsychotic medications, RisperdalÂ® ConstaÂ® versus AbilifyÂ®, over a 2-year treatment period in the long-term maintenance of patients with schizophrenia.

DETAILED DESCRIPTION:
Although many patients with schizophrenia currently take oral antipsychotic medications, it is estimated that up to 75% of them have difficulty adhering to the daily oral regimen. Long-acting injectable formulations of antipsychotics may eliminate the need for daily medication and enhance patient compliance with the treatment regimen. The purpose of this trial is to evaluate the long-term effectiveness of Risperdal® Consta®, a long-acting injectable antipsychotic medication, versus Abilify®, an oral antipsychotic medication in patients with schizophrenia. The study will include patients, who in the investigator's opinion may benefit from a change in their current antipsychotic medication due to insufficient effectiveness, side effects or difficulty in adhering to a daily dose regimen. This is an open-label, randomized study in which patients will have an equal chance of receiving treatment for up to 2 years with Risperdal® Consta®, administered in the muscles near the hip every 2 weeks, or Abilify®, taken orally once daily. The initial dose and subsequent dose of study drug will be determined by the investigator. The patient's current oral antipsychotic medication will be decreased over the first four weeks of the study and discontinued. During the study, investigators may adjust the dose of study drug or add new antipsychotic medications to treat worsening psychotic symptoms. Patients may continue on or have added, antidepressants, mood stabilizers (except carbamazepine), sedative hypnotics, or anxiolytic medications during the study. Patients will return to the doctor's office every two weeks to receive an injection of Risperdal® Consta® or another supply of Abilify®. During certain visits, patients will be asked questions which will help the investigator determine the severity of the patient's illness, how well the study drug is working, quality of life, reasoning, memory, judgement and perception and side effects that may be associated with schizophrenia or treatment. Safety evaluations include the incidence of adverse events during the study, vital signs and clinical laboratory tests (both blood and urine). The study hypothesis is that Risperdal® Consta® is superior to Abilify® in the long-term treatment of subjects with schizophrenia as measured by time to relapse and time in remission. Treatment with Risperdal® Consta® (administered in the muscle every 2 weeks) at a dose of 25, 37.5 or 50 mg or Abilify® (administered orally daily) at a dose of 10-30 mg for 2 years. Investigators will determine the starting dose and may adjust the dosage of study drug during the study according to symptoms and treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of schizophrenia
* Patient has had at least 2 psychotic relapses in the two years prior to study entry
* patient is not adequately benefiting from their current antipsychotic medication

Exclusion Criteria:

* Patients that have been hospitalized or had major medication changes within 2 months of study entry
* Patients currently experiencing, or who have experienced worsening of disease symptoms within 2 months of study entry
* Patients currently using clozapine or carbamazepine
* Patients who have undergone electroconvulsive therapy or depot antipsychotic treatment within 6 months prior to study entry
* pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2006-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient in was on February 28, 2006; last patient out was on January 26, 2009. Enrollment occurred across multiple sites in the United States, Argentina, Chile, and India and patients were enrolled from outpatient psychiatric clinics associated with private medical practices, private clinical trial sites, and academic medical centers.
Pre-assignment Details: A Screening Visit (maximum of 14 days) prior to the Treatment Phase. Baseline included psychiatric exam, lab, ECG, and schizophrenia symptom rating scale. Subjects were permitted to remain on previous psychotropic medications (i.e., antipsychotic, antidepressant, mood stabilizer, anxiolytics) up to the first 4 weeks of the Treatment Phase.
Groups:
- Risperdal Consta: 25mg, 37.5mg, or 50mg every 2 weeks injection for 104 weeks
- Abilify: 10-30 mg once daily oral for 104 weeks
Period: Overall Study
Arm/Group | Risperdal Consta | Abilify
Started | 179 | 176
Completed | 126 | 126
Not Completed | 53 | 50
Not completed — Death | 1 | 0
Not completed — Adverse Event | 0 | 4
Not completed — Lost to Follow-up | 18 | 10
Not completed — Withdrawal by Subject | 25 | 23
Not completed — Pregnancy | 0 | 1
Not completed — Insufficient Response | 4 | 3
Not completed — Admin issues, sponsor decision, etc. | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Risperdal Consta | Abilify | Total
Number analyzed (Participants) | 179 | 176 | 355
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 177 | 173 | 350
  >=65 years | 2 | 3 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 38.3 (11.66) | 37.8 (11.49) | 38 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 70 | 143
  Male | 106 | 106 | 212
Region of Enrollment [Number; unit: participants]
  India | 91 | 91 | 182
  United States | 51 | 52 | 103
  South America | 37 | 33 | 70

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse
Description: Time to relapse was defined as the number of days from the date of first dose to the date of relapse, as determined by the Relapse Monitoring Board.
Time Frame: Day 1 to relapse
Population: explanatory ITT analysis data set (eITT) contains all subjects who had at least one administration of study drug as well as at least one follow-up efficacy measurement; includes assessments while the subject is on study drug.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Risperdal Consta | Abilify
Number analyzed (Participants) | 177 | 172
days | 131 [100 to 197] | 113 [99 to 169]
Statistical Analysis 1: Comparison: Risperdal Consta vs Abilify; Null hypothesis: there is no difference in time to relapse; Test type: Superiority or Other; p = 0.684, Log Rank — Hochberg procedure was used for adjusting multiple endpoint comparisons; Insufficient number of subjects who had an event for median estimation

2. Primary Outcome: Time in Remission
Description: Time in remission for an individual subject was defined as the length of time (in days) that the remission criteria were maintained during the trial. Remission was defined as the simultaneous attainment of a score of 3 (mild), 2 (minimal), or 1 (absent) for all the following individual items from Positive and Negative Syndrome Scale (PANSS): delusions (P1), concept disorganization (P2), hallucinatory behavior (P3), unusual thought content (G9), mannerisms and posturing (G5), blunted affect (N1), passive/apathetic social withdrawal (N4), and lack of spontaneity and flow of conversation (N6).
Time Frame: Day 1 to last PANSS measurement
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Risperdal Consta | Abilify
Number analyzed (Participants) | 179 | 176
days | 373.5 (282.6) | 356.7 (291.99)
Statistical Analysis 1: Comparison: Risperdal Consta vs Abilify; Null hypothesis: there is no difference in time in remission between the two treatment groups; Test type: Superiority or Other; p = 0.646, Wilcoxon (Mann-Whitney) — Hochberg procedure was used for adjusting multiple endpoint comparisons

ADVERSE EVENTS:
Time Frame: Adverse events were reported as treatment emergent if the onset date is before or within 49 days of last dose of RISPERDAL CONSTA or before or within 30 days of last dose of Abilify.
Arm/Group | RISPERDAL CONSTA | Abilify
Serious Adverse Events (participants affected / at risk) | 31/179 | 35/176
Other Adverse Events (participants affected / at risk) | 151/179 | 141/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RISPERDAL CONSTA (N=179) | Abilify (N=176)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 | 0
GOITRE (Endocrine disorders) | 0 | 1
ANAL FISSURE (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 1
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 0 | 1
MELAENA (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1
DEATH (General disorders) | 1 | 0
PYREXIA (General disorders) | 0 | 1
CELLULITIS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 1
MULTIPLE DRUG OVERDOSE ACCIDENTAL (Injury, poisoning and procedural complications) | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
AKATHISIA (Nervous system disorders) | 1 | 0
CONVULSION (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 0 | 1
PSYCHOTIC DISORDER (Psychiatric disorders) | 12 | 11
SCHIZOPHRENIA (Psychiatric disorders) | 7 | 12
SUICIDAL IDEATION (Psychiatric disorders) | 2 | 1
AGGRESSION (Psychiatric disorders) | 2 | 0
DEPRESSION SUICIDAL (Psychiatric disorders) | 2 | 0
AFFECT LABILITY (Psychiatric disorders) | 1 | 0
ALCOHOLISM (Psychiatric disorders) | 0 | 1
ANXIETY (Psychiatric disorders) | 0 | 1
COMPLETED SUICIDE (Psychiatric disorders) | 0 | 1
DRUG DEPENDENCE (Psychiatric disorders) | 0 | 1
HOMICIDAL IDEATION (Psychiatric disorders) | 1 | 0
MANIA (Psychiatric disorders) | 0 | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RISPERDAL CONSTA (N=179) | Abilify (N=176)
HYPERPROLACTINAEMIA (Endocrine disorders) | 9 | 0
DIARRHOEA (Gastrointestinal disorders) | 12 | 19
VOMITING (Gastrointestinal disorders) | 18 | 13
NAUSEA (Gastrointestinal disorders) | 16 | 11
CONSTIPATION (Gastrointestinal disorders) | 14 | 12
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 6 | 11
SALIVARY HYPERSECRETION (Gastrointestinal disorders) | 7 | 9
PYREXIA (General disorders) | 26 | 21
FATIGUE (General disorders) | 10 | 17
ASTHENIA (General disorders) | 7 | 14
INJECTION SITE PAIN (General disorders) | 9 | 1
NASOPHARYNGITIS (Infections and infestations) | 18 | 16
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 | 18
INFLUENZA (Infections and infestations) | 11 | 7
WEIGHT INCREASED (Investigations) | 15 | 15
DECREASED APPETITE (Metabolism and nutrition disorders) | 29 | 16
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 14 | 14
BACK PAIN (Musculoskeletal and connective tissue disorders) | 12 | 14
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 12 | 12
TREMOR (Nervous system disorders) | 39 | 40
HEADACHE (Nervous system disorders) | 30 | 27
AKATHISIA (Nervous system disorders) | 20 | 20
DIZZINESS (Nervous system disorders) | 25 | 13
HYPERSOMNIA (Nervous system disorders) | 11 | 10
SOMNOLENCE (Nervous system disorders) | 12 | 7
SEDATION (Nervous system disorders) | 10 | 6
INSOMNIA (Psychiatric disorders) | 47 | 51
PSYCHOTIC DISORDER (Psychiatric disorders) | 30 | 30
ANXIETY (Psychiatric disorders) | 32 | 26
SCHIZOPHRENIA (Psychiatric disorders) | 25 | 21
DEPRESSION (Psychiatric disorders) | 24 | 15
RESTLESSNESS (Psychiatric disorders) | 11 | 5
SLEEP DISORDER (Psychiatric disorders) | 7 | 9
COUGH (Respiratory, thoracic and mediastinal disorders) | 17 | 12

LIMITATIONS AND CAVEATS:
15% of subjects did not meet stability inclusion criteria; many received supplemental antipsychotics post-randomization; biweekly visits may have increased aripiprazole adherence; numerous early dropouts may have led to dependent censoring and bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less